CLINICAL TRIAL: NCT01308242
Title: Effects of a Non-Calcium Based Phosphate Binder on FGF23 Levels in Chronic Kidney Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 33139CS
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Patients enrolled will receive Renvela for a 3 month time frame.
  Interventions: Drug: Sevelamer Carbonate

INTERVENTIONS:
Drug: Sevelamer Carbonate — Sevelamer 800 mg by mouth three times daily with meals for 3 months
  Other Names: Renvela

SUMMARY:
Fibroblast Growth Factor 23 (FGF23) is a molecule that has been implicated in the homeostasis of phosphorus. Elevated FGF23 levels are well-documented in patients with Chronic Kidney Disease (CKD) and are inversely correlated with Glomerular Filtration Rate (GFR). FGF23 levels are also predictive of progression of CKD and predict mortality in CKD. Although studies in normal individuals suggest that phosphorus intake is related to FGF23 levels, the effect of dietary and pharmacologic phosphate restriction on FGF23 levels in patients with CKD has never been reported. Our objectives are to determine if phosphate reduction through the use of non-calcium based phosphate binder will decrease serum FGF23 levels. The investigators will also be investigating associations of elevation in FGF 23 levels with commonly encountered co-morbidities in CKD patients such as Coronary Artery Disease, Diabetes Mellitus, and Hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults between ages 18-80 years old, with a GFR less than or equal to 50 ml/min/1.73 m2 as determined by the Modification of Diet in Renal Disease (MDRD) formula will be included.

Exclusion Criteria:

* Patients will be excluded if they have a history of renal transplant or are pregnant. In addition, patients with dysphagia, swallowing disorders, severe GI motility disorders, severe constipation, history of major gastrointestinal surgery and patients taking levothyroxine for hypothyroidism will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

PRIMARY OUTCOMES:
Effects of a Non-Calcium Based Phosphate Binder on FGF23 Levels in Chronic Kidney Disease | March 2011-June 2012
  Determine if phosphate reduction through the use of non-calcium based phosphate binders will decrease serum FGF23 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States